CLINICAL TRIAL: NCT02436252
Title: Phase 1/2 Study of DSP-7888 in Patients With Myelodysplastic Syndrome (MDS)
Brief Title: Study of DSP-7888 in Patients With Myelodysplastic Syndrome
Acronym: MDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DB650027
Record Dates: First submitted 2015-04-23; First posted 2015-05-06 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes

ARMS (1):
- DSP-7888 (Experimental)
  Interventions: Drug: DSP-7888

INTERVENTIONS:
Drug: DSP-7888 — 3.5-10.5 mg/body,Id every 2-4 weeks

SUMMARY:
This is a phase 1/2, uncontrolled, open-label, multicenter study in patients with MDS for whom no effective therapies currently exist.

DETAILED DESCRIPTION:
This is a phase 1/2, uncontrolled, open-label, multicenter study in patients with MDS for whom no effective therapies currently exist. In the Phase 1 part, high risk and low risk patients with MDS requiring additional treatment will be enrolled, and two different dose levels of DSP-7888 (3.5 and 10.5 mg/body) will be investigated in a stepwise manner starting with the lower dose using the 3+3 design, to determine the MTD and the RD for the Phase 2 part based on DLT evaluation during the 29 days following the initial dose of DSP-7888. In the Phase 2 part, DSP-7888 therapy at the RD determined by the Phase 1 part will be administered to high risk patients with MDS who had received and not responded to azacitidine as a standard treatment.

ELIGIBILITY:
Inclusion Criteria:

[For Phase 1 part only]

* Patients with a diagnosis of MDS according to either the fourth edition of the WHO classification or the FAB classification, with the exception of those with chronic myelomonocytic leukemia (CMML) or refractory anemia with excess blasts in transformation (RAEB-t)
* Patients with an International Prognostic Scoring System (IPSS) score of ≧ 1.5 at enrollment, or patients with an IPSS score of < 1.5 who require additional treatment to supportive therapy in the opinion of the investigator or subinvestigator.
* Patients who will be able to be hospitalized from the initial dose of DSP-7888 until the end of the post-initial dose observation (Patients may be permitted to have a temporary overnight leave during the hospitalization.)

[For Phase 2 part only]

* Patients with a diagnosis of MDS according to either the fourth edition of the WHO classification or the FAB classification
* Patients with an IPSS score of ≧ 1.5 at enrollment, or patients with an IPSS score of < 1.5 with myeloblasts ≧ 5%
* Patients who received at least one cycle of azacitidine therapy

[For both Phase 1 and 2 parts]

* Patients with a peripheral white blood cell count of ≦12,000/mm3 within 4 weeks (28 days) before enrollment (on the basis of the most recent data during the period if multiple data are available)
* Patients aged ≧20 years at the time of informed consent
* Patients who have provided written voluntary consent in person to participate in this study after fully receiving and understanding the information about this study, including study objectives, contents, expected pharmacological actions and effects, and foreseeable risks
* Patients with an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 2 at enrollment
* Patients with a life expectancy of ≧ 3 months (90 days)
* Patients for whom no standard therapies are currently available, including transplant treatments such as allogeneic stem cell transplant
* Patients with a human leukocyte antigen (HLA) type of HLA-A*24:02 or HLA-A*02:01/06
* Patients with adequate major organ functions meeting the following criteria on the basis of laboratory data within 4 weeks (28 days) before enrollment (if multiple data are available, most recent data during the period)

  * Serum creatinine: ≦ 2-fold the upper limit of the normal range of the study site (ULN)
  * Total bilirubin: ≦2-fold the ULN
  * AST, ALT: ≦3-fold the ULN
* Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to use appropriate contraception from the time of consent until 6 months (180 days) after the last dose of the study drug to avoid pregnancy
* Female patients of childbearing potential must have a negative pregnancy test (urine) within 4 weeks (28 days) before enrollment

Exclusion Criteria:

* Patients with a dry tap on bone marrow aspiration before enrollment
* Patients with grade ≧ 3 infection according to the Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE v4.0)
* Patients with a positive test result for HIV antibody, HBs antigen or HCV antibody
* Patients with any intracranial metastasis that is symptomatic or requires treatment
* Patients with active multiple cancers (synchronous multiple cancers, or metachronous multiple cancers with a disease-free period of ≦ 5 years, with the exception of carcinoma in situ, mucosal carcinoma, or other such carcinomas curatively treated with local therapy)
* Patients who had myocardial infarction within 6 months (180 days) before enrollment
* Patients with significant diseases at enrollment that may affect study treatment, such as New York Heart Association (NYHA) Functional Class III or IV heart disease, CTCAE v4.0 grade ≧ 3 arrhythmia, angina pectoris, abnormal electrocardiogram findings, interstitial pneumonia or pulmonary fibrosis
* Patients with uncontrollable complications
* Patients with CTCAE v4.0 grade ≧2 hemorrhage
* Patients who underwent allogeneic hematopoietic stem cell transplant
* Patients who received any of the following treatments within the specified period before enrollment:

  * Surgery, radiotherapy, chemotherapy (including molecular-targeted drugs): 4 weeks (28 days)
  * Immunosuppressants, cytokine preparations (excluding G-CSF): 4 weeks (28 days)
  * Endocrine therapy, immunotherapy (including biological response modifier therapy): 2 weeks (14 days)
* Pregnant women or breastfeeding women
* Patients with concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease, or patients who require long-term systemic steroid therapy (excluding therapy given on a PRN basis)
* Patients with any ongoing CTCAE v4.0 grade ≧ 2 adverse effects of prior treatment (excluding alopecia and phlebitis)
* Patients who received any investigational product or post-marketing study drug within 4 weeks (28 days) before enrollment
* Patients with a history of allergy to any oily drug products
* Patients who previously received DSP-7888, any other WT1 peptide, or WT1 immunotherapy
* Patients who are inappropriate for participation in the study for other reasons in the opinion of the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by adverse events (AEs), serious adverse events (SAEs), dose-limiting toxicity (DLT) | 12 months
  Safety and tolerability assessed by adverse events (AEs), serious adverse events (SAEs), dose-limiting toxicity (DLT)
Overall Survival （OS） | 24 months
  Participants follow-up for overall survival will occur. Maximum follow-up time is 2 year after the initial administration of the last subject.

SECONDARY OUTCOMES:
Overall Response Rate（ORR） | 6 months
  HR（Hematologic Response）, HI（Hematologic improvement） and Cytogenetic response assessed by IWG MDS response criteria 2006
TI （Blood transfusion independence） | 6 months
  Defined as the absence of any RBC or PLT transfusion for any consecutive 8 weeks
Time to transformation to AML | 24 months
  Participants follow-up for time to transformation to AML will occur. Maximum follow-up time is 2 year after the initial administration of the last subject.
Biomarkers | 6 months
  Explore efficacy related biomarkers assessed by delayed-type hypersensitivity (DTH) reactions to WT1 peptide and WT1 peptide-specific CTL-induction activity

CONTACTS AND LOCATIONS:
Overall Officials: Sumitomo Pharma Co., Ltd. Japan, Study Director — Sumitomo Pharma Co., Ltd.
Locations (16):
- Japan (16):
  - Japanese Red Cross Narita Hospital, Narita, Chiba
  - Chugoku Central Hospital, Fukuyama, Hiroshima
  - Yokohama Municipal Citizen's Hospital, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Sendai Medical Center, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Tokyo Metropolitan Geriatric Hospital, Itabashi-ku, Tokyo
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Okayama City General Medical Center Okayama City Hospital, Okayama